CLINICAL TRIAL: NCT00149123
Title: Low-dose Hydrocortisone in the Treatment of the Shock of Burned Patients
Brief Title: Low-dose Hydrocortisone in Acutely Burned Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 2004.354
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2007-10

CONDITIONS: Burns
Keywords: Burn; adrenal insufficiency; hydrocortisone; short corticotropin test
MeSH Terms: conditions — Burns; Adrenal Insufficiency | interventions — Hydrocortisone

INTERVENTIONS:
Drug: hydrocortisone 200 mg/day

SUMMARY:
Major burns trigger the release of circulating mediators, as cytokines and endotoxin that induces a systemic inflammatory response syndrome. The cardiovascular effects are similar to those seen in septic shock. After the initial hypovolemic phase, patients with extensive burns often present a shock with increased cardiac output and reduced systemic vascular resistances. As described in septic shock, we test the hypothesis that low-dose hydrocortisone could decrease the duration of the shock period.

ELIGIBILITY:
Inclusion Criteria:

* males and females,
* between 18 and 75 year old
* who present a burned surface more than 30% of the body surface
* who need catecholamine infusion
* between J0 and J3 after the injury.

Exclusion Criteria:

* pregnancy,
* trauma,
* sepsis,
* cardiac insufficiency,
* AIDS,
* etomidate administration

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-04; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Number of patients who do not receive any more catecholamine 4 days after the beginning of the shock

SECONDARY OUTCOMES:
Duration of catecholamine administration
Doses of administered catecholamine
Adrenal insufficiency incidence

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie TISSOT, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Sylvie TISSOT, Lyon, France

REFERENCES:
- [Derived] Plassais J, Venet F, Cazalis MA, Le Quang D, Pachot A, Monneret G, Tissot S, Textoris J. Transcriptome modulation by hydrocortisone in severe burn shock: ancillary analysis of a prospective randomized trial. Crit Care. 2017 Jun 16;21(1):158. doi: 10.1186/s13054-017-1743-9. PMID 28623938
- [Derived] Venet F, Plassais J, Textoris J, Cazalis MA, Pachot A, Bertin-Maghit M, Magnin C, Rimmele T, Monneret G, Tissot S. Low-dose hydrocortisone reduces norepinephrine duration in severe burn patients: a randomized clinical trial. Crit Care. 2015 Jan 26;19(1):21. doi: 10.1186/s13054-015-0740-0. PMID 25619170